CLINICAL TRIAL: NCT03698253
Title: Prognostic Value of EGFR Expression, KRAS Mutation and Tumor Sideness in Patients With Metastatic Colorectal Cancer Treated With Regorafenib and FOLFIRI as a Third- or Fourth-line Setting
Brief Title: Metastatic Colorectal Cancer Treated With Regorafenib and FOLFIRI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kaohsiung Medical University Chung-Ho Memorial Hospital (Other)
Responsible Party: Principal Investigator, Jaw-Yuan Wang, MD, PhD, Professor, Vice Superintendent, Kaohsiung Medical University Chung-Ho Memorial Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KMUHIRB-E(I)-20180270
Record Dates: First submitted 2018-10-01; First posted 2018-10-05 (Actual); Last update posted 2018-10-05 (Actual); Status verified 2018-10

CONDITIONS: Colorectal Cancer
Keywords: EGFR; KRAS; tumor sideness; FOLFIRI; regorafenib; metastatic colorectal cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — regorafenib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Regorafenib plus FOLFIRI (Experimental): Regimen for treatment consists of irinotecan (180 mg/m2 as a 120-min IV infusion for UGT1A1 genotyping (TA6/TA6) and UGT1A1 genotyping (TA6/TA7); 120 mg/m2 as a 120-min IV infusion for UGT1A1 genotyping (TA7/TA7)), followedby Leucovorin (400 mg/m2 IV infusion over 2 hours), and 5-FU (2800 mg/m2 IV infusion over a 46-hour period), repeated every 2 weeks.
  After every 2 cycles of each different dose of irinotecan, if adverse events (AEs) are under the grade 2, we will escalate the dose of 30 mg/m2. The estimated maximal dose of irinotecan is 260 mg/m2 for UGT1A1 genotyping (TA6/TA6); 240 mg/m2 for UGT1A1 genotyping (TA6/TA7); 180 mg/m2 for UGT1A1 genotyping (TA7/TA7).
  Regorafenib is administered at adjusted doseage of 120 mg daily for 3 weeks in a 4-week cycle.
  Interventions: Drug: Regorafenib; Genetic: UGT1A1 genotyping (TA6/TA6); Genetic: UGT1A1 genotyping (TA6/TA7); Genetic: UGT1A1 genotyping (TA7/TA7)

INTERVENTIONS:
Drug: Regorafenib — Regorafenib is administered at dose of 120 mg daily for 3 weeks in a 4-week cycle
  Other Names: stivarga
Genetic: UGT1A1 genotyping (TA6/TA6) — The dosage of irinotecan in FOLFIRI is escalated from 180mg/m2 to 260 mg/m2
Genetic: UGT1A1 genotyping (TA6/TA7) — The dosage of irinotecan in FOLFIRI is escalated from 180mg/m2 to 240 mg/m2
Genetic: UGT1A1 genotyping (TA7/TA7) — The dosage of irinotecan in FOLFIRI is escalated from 120mg/m2 to180 mg/m2

SUMMARY:
The survey is a retrospective study to evaluate the prognotic value of EGFR expression, KRAS mutations and tumor sideness in patients with metastatic colorectal cancer treated with regorafenib and FOLFIRI as a third- or fourth-line setting.

DETAILED DESCRIPTION:
Primary objective:

Progression-free survival

Secondary objecive:

Overall survival, best objective response, disease control rate and adverse events

Number of Subjects: 41 patients with metastatic colorectal cancer treated with regorafenib and FOLFIRI as a third- or fourth-line setting.

Plan of the Study:

1. This is a retrospective study.
2. Study Schedule Study date: the time getting approval letter issued by both regulatory authority and institutional review board (IRB). Duration of the study: 5 years.
3. Duration of Treatment: Treatment was administered until disease progressed.

ELIGIBILITY:
Inclusion Criteria:

* Age between 20-85 years old
* Histologically proven metastatic colorectal cancer (mCRC).
* Patients with progressing mCRC who were previously treated with FOLFOX, FOLFIRI, anti-VGFR monoclonal antibody (MoAb), and anti-EGFR MoAb if KRAS-wild-type tumors were identified.
* Patient was able to understand the requirements of the study and written informed consent was obtained from each subject.

Exclusion Criteria:

* Patients who do not meet the including criteria or unwilling to participate

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2013-10-01 (Actual); Primary Completion 2018-06-01 (Actual); Study Completion 2018-06-01 (Actual)

PRIMARY OUTCOMES:
Progression-free survival | From date of initiaton of treatment until the date of first documented progression, assessed up to 23 months
  Time from treatment to disease progresses

SECONDARY OUTCOMES:
Overall survival | From date of initiation of treatment until the date of death from any cause, assessed up to 23 months
  Time from treatment to death of subjectives
Best objective response | From date of initiation of treatment until the date of disease progression, assessed up to 23 months
  best response recorded during treatment
Disease control rate | From date of initiation of treatment until the date of disease progression, assessed up to 23 months
  Rate of best objective response, including complete response, partial response and stabel disease
Rate of treatment-associated adverse events. | Adverse events is evaluated and recorded during every cycle of treatment. Up to 23 months.
  Common Terminology Criteria for Adverse Events version 3.0 was used for evaluating treatment-associated adverse events.

CONTACTS AND LOCATIONS:
Overall Officials: Jaw-Yuan Wang, PhD, Study Chair — Division of Colorectal Surgery, Department of Surgery, Kaohsiung Medical University Hospital, Kaohsiung Medical University
Locations (1):
- Chung-Ho Memorial Hospital, Kaohsiung Medical University:, Kaohsiung City, Taiwan

IPD SHARING:
Plan to Share IPD: No